CLINICAL TRIAL: NCT04854343
Title: SLPI: a Novel Biomarker of Prostate Cancer
Brief Title: SLPI for Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Florence (Other)
Collaborators: Istituto per lo Studio, la Prevenzione e la Rete Oncologica (Other); Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Simone Morselli, PhD Student, University of Florence
Other Study IDs: 17931
Record Dates: First submitted 2021-04-13; First posted 2021-04-22 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Prostate Cancer; Prostatic Neoplasm
Keywords: Prostate; SLPI; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Case: 200 patients with a suspicion of prostate cancer
  Interventions: Diagnostic Test: Secretory leukocyte protease inhibitor (SLPI) in prostate cancer; Diagnostic Test: Determination of molecular alterations
- Control A: (a) 50 patients with benign prostate hyperplasia (BPH)
  Interventions: Diagnostic Test: Determination of molecular alterations; Diagnostic Test: Secretory leukocyte protease inhibitor (SLPI) Healthy
- Control B: (b) 30 male subjects older than 50 years with neither prostate disease nor any other neoplasia
  Interventions: Diagnostic Test: Secretory leukocyte protease inhibitor (SLPI) Healthy

INTERVENTIONS:
Diagnostic Test: Secretory leukocyte protease inhibitor (SLPI) in prostate cancer — 7 ml of peripheral blood and a urine sample for the determination of SLPI concentration. Blood samples will be promptly processed to obtain sera; both sera and urine will be stored at -80°C in the laboratory. The levels of SLPI in the serum and in the urine will be quantitated by an ELISA assay by using the "Human SLPI Quantikine ELISA Kit". SLPI level will be measured at diagnosis and during the follow-up (3, 9, 15 months and in case of progression).
  Immunohistochemistry protocol for SLPI immunostaining to investigate SLPI levels prostate tissue
  Groups: Case
Diagnostic Test: Determination of molecular alterations — The presence of ETS translocation (or of ETS overexpression) will be tested on bioptic samples in each patient as for routine diagnostic procedures. First, ERG overexpression will be investigated by ERG immunostaining. The samples negative for ERG immunostaining will be studied for TMPRSS2-ERG translocation either by in situ FISH or by a translocation-specific RT-PCR. Next, the biopsies negative for TMPRSS2-ERG will be tested for the overexpression of other ETS proteins (ETV1, ETV4, ETV5 and for others rarely occurring ETS). When possible, it will be determined the status of pTEN gene, the tumor suppressor most frequently lost in prostate patients. The patients negative for the overexpression of the ETS proteins will be tested for SPINK1.
  Groups: Case; Control A
Diagnostic Test: Secretory leukocyte protease inhibitor (SLPI) Healthy — SLPI level will be measured also in the serum and in the urine from controls (patients with BPH and healthy subjects).
  7 ml of peripheral blood and a urine sample for the determination of SLPI concentration. Blood samples will be promptly processed to obtain sera; both sera and urine will be stored at -80°C in the laboratory. The levels of SLPI in the serum and in the urine will be quantitated by an ELISA assay by using the "Human SLPI Quantikine ELISA Kit".
  Groups: Control A; Control B

SUMMARY:
Exploratory study of SLPI expression in human prostate cancer patients This is a no-profit exploratory study about the expression of SLPI in human prostate cancer patients that will enroll about 200 patients admitted for suspect prostate cancer to Careggi University Hospital. We will verify whether an increase SLPI levels in the sera may serve as biomarker of cancer progression.

DETAILED DESCRIPTION:
Prostate cancer (PC) is a heterogeneous disease that occurs more frequently in elderly men. Prostate cancer is usually localized and it has a slow progression; thus, the patient may not suffer from any symptom for years. However, a proportion of patients PC develops metastases and may become a clinically relevant disease that can show an aggressive behavior and, eventually, give metastases. In any event, since it is the most common male cancer in the Western countries, it is the second leading cause of cancer deaths in males. For this reason the identification of the molecular alterations determining the different clinical behaviors and of the associated biomarkers would be extremely useful.

The Secretory leukocyte protease inhibitor (SLPI) is a serine protease which best-defined function is to protect host tissues from the excessive damage by proteolytic enzymes released during inflammation. Recently SLPI has been found overexpressed in a variety of cancers (pancreatic, papillary thyroid, uterine cervix, endometrial, and ovarian cancer). In apparent contrast, SLPI has been found reduced in the sera (and tumor tissue) of prostate cancer patients in the respect of healthy subjects and of subjects with benign hyperplasia. However, SLPI has been found upregulated in castration resistant prostate cancer (CRPC) patients and in a subset of CRPC cell lines.

These data suggest that expression of SLPI in prostate cancer could be biphasic: underexpressed during the early stages and overexpressed during progression. This peculiar pattern of SLPI expression suggests that SLPI may play a role in prostate cancer pathogenesis and/or in determining its neoplastic features. In this respect, it is noteworthy that SLPI is located at 20q13.2 (HPC20 locus), a locus harboring prostate cancer susceptibility genes. Based on these data it is possible to hypothesize that prostate cancer progression could be associated, and possibly heralded, by the increase of SLPI.

This is an observational investigation of SLPI levels in blood and tissue samples of patients with prostate disease with the explorative goal to verify whether SLPI could be a potential biomarker of prostate cancer progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prostate carcinoma.
* Patients with Benign Prostatic Hyperplasia.
* Male subjects older that 50 years without prostate or neoplastic diseases.

Exclusion Criteria:

* Male subjects younger that 50 years without prostate disease.
* Male subjects with neoplastic diseases either than prostate.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This study will be enroll patient with prostate carcinoma and, as control groups, patients with benign prostate hyperplasia (BPH) and males older than 50 years with neither prostate disease nor any other neoplasia.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
SLPI and Clinical data | through study completion, at least 15 months
  Correlation between clinical data of prostate cancer and SLPI levels
SLPI and Pathological data | Enrollment
  Correlation between pathological data of prostate cancer and SLPI levels
SLPI and Molecular Features | Enrollment
  Correlation between molecular features of prostate cancer and SLPI levels

CONTACTS AND LOCATIONS:
Overall Officials: Rosario Notaro, MD, Principal Investigator — ISPRO
Locations (1):
- Careggi University Hospital, Florence, Tuscany, Italy